CLINICAL TRIAL: NCT04999904
Title: A Proprioceptive Training Program Using an Uneven Terrain Treadmill for Patients With Ankle Instability
Acronym: ROCKY REHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Fort Sam Houston (Unknown); Naval Hospital Camp Pendleton (U.S. Federal Agency); Naval Health Research Center (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 937017; W81XWH-20-2-0056 (Other Grant/Funding Number: Congressionally Directed Medical Research Program (CDMRP): Peer Reviewed Orthopedic Research Program (PRORP))
Record Dates: First submitted 2021-07-20; First posted 2021-08-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Instability; Ankle (Ligaments) (Old Injury); Sprain of Ankle
Keywords: Acute Ankle Sprain; Chronic Ankle Instability; Proprioceptive Training; Uneven Treadmill; Reinjury; Rehabilitation; Service Members
MeSH Terms: conditions — Ankle Injuries; Reinjuries

STUDY DESIGN:
Intervention Model Description: The study will be implemented using multi-site, parallel randomized clinical trial. Individuals will be randomly allocated between a control and experimental arm, stratified between lateral ankle sprains and chronic ankle instability.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uneven Treadmill Arm (Experimental): Uneven Treadmill Intervention with up to twelve sessions over approximately six weeks and Standard of Care Physical Therapy with an 18 month follow-up period
  Interventions: Other: Uneven Treadmill Intervention
- Control Arm (Active Comparator): Standard of Care Physical Therapy over approximately six weeks with an 18 month follow-up period
  Interventions: Other: Standard of Care Physical Therapy

INTERVENTIONS:
Other: Uneven Treadmill Intervention — Progressive proprioceptive training on the uneven treadmill with up to twelve training sessions. Subjects will be advanced through activities with progression pragmatically assessed by the physical therapists for the benefit and tolerance of the individual subject. Activities may include: slow walking, fast walking, inclined/declined walking, head turning, vision obstruction, dual task walking, fatigued walking, load carriage. Standard of care physical therapy is still provided.
  Arms: Uneven Treadmill Arm
Other: Standard of Care Physical Therapy — Standard of Care Physical Therapy
  Arms: Control Arm

SUMMARY:
The ROCKY REHAB trial will provide a pragmatic approach to evaluate if incorporating a rocky, uneven terrain treadmill into the proprioceptive rehabilitation received during physical therapy can improve outcomes and reduce reinjury rates in patients with ankle instability.

DETAILED DESCRIPTION:
Lower limb sprains and strains are three-times more prevalent than any other acute injury in the Armed Forces, with lateral ankle sprains being the most common injury sustained during active-duty. Many individuals who experience an ankle sprain will go on to develop chronic ankle instability. Training and rehabilitation programs that incorporate proprioceptive training are particularly effective at improving outcomes and reducing re-injury rate. However, current programs do not help individuals "train to the tasks" that will be encountered once those individuals leave physical therapy. The proposed intervention evaluates the use of a rocky, uneven terrain treadmill that specifically targets aspects of the real-world environment for restoring and improving short-term function and performance and reducing the long-term risk of re-injury. This trial will randomly allocate 312 individuals with ankle sprains and chronic ankle instability to standard of care physical therapy or the standard of care supplemented with the uneven treadmill intervention. Patient reported outcome, performance measures, and biomechanical measures of muscle activations and plantar pressures will be evaluated. Patient reported outcomes and reinjury rates will be tracked for 18 months.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18-49.
2. Score < 24 on the Cumberland Ankle Instability Tool.
3. Foot and Ankle Ability Measure Activities of Daily Living score ≤ 90 and Sports score ≤ 80 indicating substantial ankle-foot impairment and activity limitation.
4. Able to attend treatment sessions for approximately a 6-week period.
5. Passed most recent physical fitness test (Active duty only).
6. Acute lateral ankle sprain specific inclusion criteria:

   1. history of a first-time ankle sprain that resulted in activity limitation that lasted at least one day.
   2. chronicity of 2-6 weeks prior to consent.
7. Chronic ankle instability specific inclusion criteria:

   1. history of at least one significant ankle sprain within the 12 months prior to enrollment that interrupted physical activity for 1+ days.
   2. most recent ankle sprain in the past 2-12 weeks.
   3. history of the previously injured ankle joint "giving way" and/or recurrent sprain and/or ''feelings of instability.''
8. Individual is about to start care with physical therapy.

Exclusion Criteria

1. Unable to walk at the point of study enrollment.
2. Non-removable casting.
3. History of previous surgeries to the musculoskeletal structures (i.e., bones, joint structures, nerves).
4. History of fracture in either limb of the lower extremity requiring realignment.
5. Acute injury to musculoskeletal structures of other joints of the lower extremity within the previous three months, which impacted joint integrity and function resulting in at least one interrupted day of physical activity.
6. Pregnant.
7. Self-reported disability due to neuromuscular impairment in the lower extremity, neurological or vestibular impairment that affected balance.
8. Connective tissue disorder (e.g. Marfan Syndrome or Ehlers-Danlos syndrome).
9. Anyone separating from the military within 12 months (other than normal military retirement), pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Cumberland Ankle Instability Tool | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Cumberland Ankle Instability Tool is a 9-item questionnaire, 30 points max score, with higher scores indicating better function. The Cumberland Ankle Instability Tool evaluates the severity of ankle instability during sport and activities of daily living, as well as pain.
Change in the Foot and Ankle Ability Measure, Activities of Daily Living Subscale | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Foot and Ankle Ability Measure: Activities of Daily Living subscale is a 21-item questionnaire with 84 points max, with higher scores indicating better function. The Activities of Daily Living Subscale is used to assess activity limitations and restrictions for individuals with foot and ankle disorders, including ankle sprains, during activities of daily living.
Change in the Foot and Ankle Ability Measure, Sports Subscale | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Foot and Ankle Ability Measure: Sports subscale is a 8-item questionnaire with 32 points max, with higher scores indicating better function. The Sports Subscale is used to assess activity limitations and restrictions for individuals with foot and ankle disorders, including ankle sprains, during recreational/sport activities.

SECONDARY OUTCOMES:
Change in the Lower Extremity Functional Scale | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Lower Extremity Functional Scale is a 20-item questionnaire with 80 points max, with higher scores indicating better function. The Lower Extremity Functional Scale is used for individuals with lower extremity musculoskeletal disorders and assesses activity limitations and participation restrictions.
Change in the Tampa Scale of Kinesiophobia | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Tampa Scale of Kinesiophobia is a 11-item questionnaire with scores between 11 and 44 points, with higher scores indicating greater kinesiophobia. The Tampa Scale of Kinesiophobia is used to assess subjective ratings of fear-related concepts.
Change in the Numeric Pain Rating Scale | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Numeric Pain Rating Scale is a 4-item questionnaire with scores between 0 and 40 points, with higher scores indicating greater pain. In the Numeric Pain Rating Scale subjects select a value that is most in line with the intensity of pain they have experienced in the past 24 hours.
Change in the Godin Leisure-Time Physical Activity Questionnaire | Baseline assessment (0 weeks), first ( 2 weeks) and second (4 weeks) interim assessments, discharge assessment (6 weeks) and follow-up assessments at 3, 6, 9, 12, 15, and 18 months.
  The Godin Leisure-Time Physical Activity Questionnaire measures the number of instances where subjects engaged in mild, moderate, and strenuous physical activity for greater than 15 minutes. Modified to account over the previous week rather than a typical week. Higher scores indicate more physical activity where 3, 5, and 9 points are given for each time a mild, moderate, or strenuous activity is engaged.
Change in the Y Balance Test | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  The Y Balance Test measures the distance a subject can reach in three directions, anterior, posteromedial and posterolateral without moving a support foot or touching the reach foot to the floor. The Y Balance Test is scored based on the composite reach distance normalized by the subject's leg length.
Change in the Side Hop Test | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  The Side Hop Test measures the how long in seconds it takes for a subject can hop on one foot across two lines spaced 30 cm apart.
Change in the Edgren Side Step Test | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  The Edgren Side Step Test measures the distance in meters a subject sidestep across in 10 seconds traversing 5 lines 1 meter apart before reversing direction.
Change in the T-Test | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  The T-Test measures the time it takes for a subject to traverse a 40m course in the shape of a "T" consisting of 10m each of forward motion, right side shuffle, left side-shuffle, and backwards motion.
Change in Electromyography (EMG) | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  EMG will be collected during walking to examine muscle activation timings and magnitudes.
Change in the Plantar Pressures | Baseline assessment (0 weeks) and discharge assessment (6 weeks).
  Plantar Pressures will be collected during walking to examine pressure distribution and progression of the center of pressure during stance phase.
Ankle Reinjury Status | Over an 18 month follow-up period.
  Timing of any ankle reinjuries during the follow-up period period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Pinata Sessoms, PhD, Principal Investigator — Naval Health Research Center
Locations (2):
- United States (2):
  - Naval Hospital Camp Pendelton, Oceanside, California
  - Naval Medical Center San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified primary outcome data will be published. Additional outcome data may also be included.
Supporting Information: Study Protocol
Time Frame: Roughly 12 months after data collection completion as part of study publications.

REFERENCES:
- [Derived] Russell Esposito E, Farrokhi S, Shuman BR, Sessoms PH, Szymanek E, Hoppes CW, Bechard L, King D, Fraser JJ. Uneven Treadmill Training for Rehabilitation of Lateral Ankle Sprains and Chronic Ankle Instability: Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 22;11(6):e38442. doi: 10.2196/38442. PMID 35731551